CLINICAL TRIAL: NCT05716672
Title: Impact of Lazertinib Dose Modification on Effectiveness and Safety in EGFR T790M-Positive Advanced Lung Cancer
Brief Title: Impact of Lazertinib Dose Modification on Effectiveness and Safety
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pusan National University Hospital (Other)
Collaborators: Yuhan Corporation (Industry)
Responsible Party: Principal Investigator, Min Ki Lee, Professor, Pusan National University Hospital
Other Study IDs: PNU-001; LASER IIT-018 (Other Grant/Funding Number: Yuhan Corporation)
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; EGFR-TKI; Lazertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lazertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 240mg group: Maintenance of the 240mg dose for 12 weeks after the first administration of Lazertinib
  Interventions: Drug: Lazertinib
- 160mg group: Reduction of the 160mg dose for 12 weeks after the first administration of Lazertinib
  Interventions: Drug: Lazertinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib 240mg(3tablets, 80mg/1tablet), once a day(QD), oral(PO), until disease progression or unacceptable toxicity
  Other Names: LECLAZA

SUMMARY:
The primary objective is to evaluate Progression Free Survival (PFS) of the group (160 mg group) in which dose reduction was performed for 12 weeks after the first administration of Lazertinib.

The Secondary objectives of this study are as follows.

1. To evaluate Progression-free survival (PFS) of the group maintaining the same dose (240mg group) and the group in which dose reduction was performed (160mg group) for 12 weeks after the first administration of Lazertinib
2. In the group maintaining the same dose (240mg group) and the group in which dose reduction was performed (160mg group) for 12 weeks after the first administration of Lazertinib, Time-to-Treatment Discontinuation(TTD), Objective Response Rate(ORR), Disease Control Rate(DCR), Tumor shrinkage and Overall Survival(OS) is evaluated.
3. In the group maintaining the same dose (240mg group) and the group in which dose reduction was performed (160mg group) for 12 weeks after the first administration of Lazertinib, specific reasons (adverse event name, grade, etc.) according to Lazertinib dose adjustment is evaluated.
4. To evaluate the treatment profile of Lazertinib including duration of treatment, dose adjustment, and reason for discontinuation of treatment.
5. To evaluate the safety of Lazertinib in the 240 mg and 160 mg groups

DETAILED DESCRIPTION:
This study is a prospective multi-center observational study, and 11 institutions will participate to enroll 200 subjects competitively. We will evaluate the efficacy and safety of Lazertinib according to maintenance of the 240mg dose and reduction of the 160mg dose for 12 weeks after the first administration of Lazertinib in non-small cell lung cancer patients confirmed to be T790M mutation-positive after treatment failure with first- or second-generation EGFR-TKIs. The study period is up to 3 years from the date of IRB approval. Follow-up is 2 years from the last subject enrollment, and data will be collected through periodic medical record review during Lazertinib administration for enrolled subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who agreed in writing to participate in this study
2. Adult men and women over 20 years of age
3. Patients with locally advanced or metastatic, recurrent non-small cell lung cancer with EGFR mutation (based on AJCC 8th edition)
4. Patients with confirmed disease progression after 1st or 2nd generation EGFR-TKI treatment
5. Patients scheduled to receive Lazertinib after T790M mutation was confirmed positive in tissue or plasma

Exclusion Criteria:

1. Patients who are receiving or have already completed Lazertinib
2. Patients whose life expectancy is less than 12 weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who agreed to participate in this study among patients scheduled to receive Lazertinib after T790M mutation was confirmed positive after treatment with 1st or 2nd generation EGFR-TKIs
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | Up to approximately 3 years
  Progression-free survival is defined as the period from the start of Lazertinib administration to the time when objective disease progression is confirmed or death from any cause during treatment, whichever occurs first.

SECONDARY OUTCOMES:
Time-to-Treatment Discontinuation (TTD) | Up to approximately 3 years
  Time-to-Treatment Discontinuation (TTD) is defined as the time from the start of Lazertinib administration to the point at which Lazertinib administration was discontinued for any reason.
Objective Response Rate(ORR) | Up to approximately 3 years
  Objective Response Rate (ORR) is defined as the proportion of subjects whose best overall response was complete response(CR) or partial response(PR) during the period of Lazertinib administration.
Disease Control Rate (DCR) | Up to approximately 3 years
  Disease Control Rate (DCR) is defined as the proportion of subjects whose best overall response was complete response(CR), partial response(PR), or stable disease(SD) during the period of Lazertinib administration.
Tumor shrinkage | Up to approximately 3 years
  Tumor shrinkage is defined as the ratio of the size of the primary lesion at the time of baseline before the first administration of Lazertinib and the size of the primary lesion at the time of maximum overall response during Lazertinib administration.
Overall Survival (OS) | Up to approximately 3 years
  Overall Survival (OS) is defined as the period from the start of Lazertinib administration to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Min Ki Lee, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (11):
- South Korea (11):
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No